CLINICAL TRIAL: NCT02024646
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Brodalumab in Subjects With Psoriatic Arthritis: AMVISION-2
Brief Title: Study of Efficacy and Safety of Brodalumab in Subjects With Psoriatic Arthritis
Acronym: AMVISION-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110144; 2013-003553-16 (EudraCT Number)
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Brodalumab; AMG 827
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 210 mg brodalumab (Experimental): Administered via subcutaneous injections.
  Interventions: Drug: 210 mg brodalumab
- 140 mg brodalumab (Experimental): Administered via subcutaneous injection.
  Interventions: Drug: 140 mg brodalumab
- Placebo (Placebo Comparator): Administered via subcutaneous injection until week 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 210 mg brodalumab — 210 mg brodalumab administered via subcutaneous injection.
  Other Names: AMG 827
  Arms: 210 mg brodalumab
Drug: 140 mg brodalumab — 140 mg brodalumab administered via subcutaneous injection.
  Other Names: AMG 827
  Arms: 140 mg brodalumab
Drug: Placebo — Placebo administered via subcutaneous injection until week 24.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of brodalumab, compared to placebo, in subjects with psoriatic arthritis. The key secondary objective is to evaluate the efficacy of brodalumab compared to placebo at week 16. The safety objective of this study is to evaluate the safety profile of brodalumab in subjects with psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

Subjects has a diagnosis of psoriatic arthritis (by the Classification of Psoriatic Arthritis criteria (CASPAR), with ≥ 3 tender and ≥ 3 swollen joints (excluding distal interphalangeal joints). Subjects must have at least

1 psoriatic skin lesion. Exclusion Criteria:

• -Subject has known history of active tuberculosis.

* Subject has a planned surgical intervention between baseline and the week 52 evaluation.
* Subject has an active infection or history of infections.
* Subject has any systemic disease (eg, renal failure, heart failure, hypertension, liver disease, diabetes, anemia) considered by the Investigator to be clinically significant and uncontrolled.
* Subject has any concurrent medical condition or electrocardiogram (ECG) abnormality that, in the opinion of the investigator, could cause this study to be detrimental to the subject.

Subject has severe depression measured by Personal Health Questionnaire Depression Scale (PHQ-8) or suicidal ideation/behavior as measured by and Columbia Suicide Severity Rating Scale (e-CSSRS)

• Subject has a history or evidence of psychiatric disorder or substance abuse considered by the Investigator to pose a risk to subject safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (83):
- United States (29):
  - Research Site, Peoria, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Cypress, California
  - Research Site, Hemet, California
  - Research Site, Huntington Beach, California
  - Research Site, La Jolla, California
  - Research Site, Palm Desert, California
  - Research Site, Palo Alto, California
  - Research Site, Victorville, California
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Paducah, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Wheaton, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Battle Creek, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Rochester, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Dallas, Texas
  - Research Site, Waco, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Seattle, Washington
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Waterloo, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
- France (7):
  - Research Site, Bordeaux
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lille
  - Research Site, Lyon Cédex 3
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Reims
- Germany (5):
  - Research Site, Frankfurt
  - Research Site, Hanover
  - Research Site, Hildesheim
  - Research Site, Leipzig
  - Research Site, Lübeck
- Greece (3):
  - Research Site, Athens
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Eger
  - Research Site, Nyíregyháza
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Szombathely
- Research Site, Riga, Latvia
- Mexico (4):
  - Research Site, Mexicali, Baja California Norte
  - Research Site, Guadalajara, Jalisco
  - Research Site, Ciudad Obregón, Sonora
  - Research Site, Mérida, Yucatán
- Poland (11):
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Stalowa Wola
  - Research Site, Świdnik
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (10):
  - Research Site, Chelyabinsk
  - Research Site, Kemerovo
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Voronezh
  - Research Site, Yekaterinburg

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Started | 163 | 160 | 161
Completed | 131 | 135 | 133
Not Completed | 32 | 25 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo | Total
Number analyzed (Participants) | 163 | 160 | 161 | 484
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [19 to 79] | 48 [22 to 80] | 49 [18 to 76] | 48 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 80 | 85 | 249
  Male | 79 | 80 | 76 | 235
Region of Enrollment [Number; unit: participants]
  Greece | 3 | 6 | 2 | 11
  Canada | 9 | 14 | 9 | 32
  Latvia | 6 | 6 | 3 | 15
  Russian Federation | 20 | 17 | 19 | 56
  Hungary | 3 | 9 | 8 | 20
  United States | 42 | 37 | 43 | 122
  Poland | 62 | 57 | 58 | 177
  Mexico | 4 | 5 | 4 | 13
  France | 7 | 2 | 2 | 11
  Germany | 7 | 7 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: ACR20 (American College of Rheumatology 20% Improvement) Response Rate Through Week 16
Description: ACR20 is used as a measurement of the proportion of subjects who are reaching a 20% improvement of tender an swollen joint counts. The higher percent of subjects reaching a higher improvement percentage shows greater success.
Time Frame: Baseline and 16 Weeks
Population: The Primary Analysis Set consists of all randomized subjects who had the opportunity to complete the week 16 visit prior to termination of the study.
  The numbers in the outcome measure data table reflect the percentage of subjects achieving ACR20.
Measure: Number; unit: Percentage of Participants
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Number analyzed (Participants) | 146 | 141 | 146
Percentage of Participants | 41.8 | 48.9 | 24.7

ADVERSE EVENTS:
Arm/Group | 210 mg Brodalumab | 140 mg Brodalumab | Placebo
Serious Adverse Events (participants affected / at risk) | 5/163 | 3/160 | 5/161
Other Adverse Events (participants affected / at risk) | 91/163 | 85/160 | 83/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 210 mg Brodalumab (N=163) | 140 mg Brodalumab (N=160) | Placebo (N=161)
ALT increased (Blood and lymphatic system disorders) | 1 | 0 | 1
Bursitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Psoriatic Arthropathy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Infection (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Abortion Induced (Surgical and medical procedures) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 2
AST Increased (Blood and lymphatic system disorders) | 0 | 0 | 1
Carotid Artery Stenosis (Vascular disorders) | 0 | 0 | 1
Cerebrovascular Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Blood and lymphatic system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 210 mg Brodalumab (N=163) | 140 mg Brodalumab (N=160) | Placebo (N=161)
Nasopharyngitis (Infections and infestations) | 28 | 17 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 16 | 16 | 2
Sinusitus (Infections and infestations) | 10 | 2 | 2
Oral Herpes (Infections and infestations) | 6 | 3 | 0
Bronchitis (Infections and infestations) | 5 | 4 | 2
Urinary Tract Infection (Infections and infestations) | 5 | 8 | 1
Pharyngitis (Infections and infestations) | 4 | 5 | 4
Influenza (Infections and infestations) | 2 | 2 | 3
Laryngitis (Infections and infestations) | 2 | 4 | 3
Herpes Zoster (Infections and infestations) | 0 | 0 | 3
Gout (Metabolism and nutrition disorders) | 5 | 0 | 0
Headache (Nervous system disorders) | 5 | 5 | 5
Hypertension (Vascular disorders) | 4 | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 6
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 13 | 6 | 4
Nausea (Gastrointestinal disorders) | 7 | 8 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 3 | 1
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 8 | 7 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 8 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4
Fatigue (General disorders) | 1 | 1 | 3
Chest Pain (General disorders) | 0 | 1 | 4
peripheral Swelling (General disorders) | 0 | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 7 | 5
Ligament Sprain (General disorders) | 4 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No